CLINICAL TRIAL: NCT02704390
Title: An Extension Study to Evaluate the Long-term Safety and Efficacy of ORADUR®-Methylphenidate in Children and Adolescents With ADHD
Brief Title: Evaluate Long-term Safety and Efficacy of ORADUR®-Methylphenidate in Children and Adolescents With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orient Pharma Co., Ltd. (Industry)
Collaborators: Durect (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OP-2PN012-301E
Record Dates: First submitted 2016-01-18; First posted 2016-03-10 (Estimated); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ORADUR®-Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ORADUR®-Methylphenidate (Experimental): ORADUR®-Methylphenidate oral capsule will be administered once daily in the morning for 24 months.
  Interventions: Drug: ORADUR®-Methylphenidate

INTERVENTIONS:
Drug: ORADUR®-Methylphenidate — ORADUR®-Methylphenidate is available in three dosage forms, 22 mg, 33 mg or 44 mg. Subjects will continue to receive ORADUR®-Methylphenidate at the previously determined optimal dose for 24 months.

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of ORADUR®-Methylphenidate in children and adolescents with ADHD.

DETAILED DESCRIPTION:
In order to evaluate the long-term safety and efficacy of ORADUR®-Methylphenidate in children and adolescents with ADHD, subjects who participated in the previous OP-2PN012-301 study will be invited to join this extension study for 24-month follow-up. Subjects will continue to receive ORADUR®-Methylphenidate at the previously determined optimal dose.

ELIGIBILITY:
Main Inclusion Criteria:

1. Subjects previously enrolled in OP-2PN012-301 study and completed 4-week study treatment
2. Both subjects and parents/guardians have provided their signed and dated informed consent form for the study

Main Exclusion Criteria:

1. Subjects who experienced unmanageable adverse events (AEs) after receiving ORADUR®-Methylphenidate
2. Subjects are taking a concomitant medication (ex: Monoamine Oxidase Inhibitor (MAOI) or other ADHD treatments) that is likely to interfere with safe administration of methylphenidate within 14 day prior to the study treatment initiation
3. Subjects are joining other clinical studies and receiving any other investigational medical products within 14 days prior to the study treatment initiation.
4. By the investigators' discretion, subjects with serious or unstable medical illness that will interfere with the evaluations of study efficacy and safety
5. By the investigators' discretion, subjects cannot understand or follow the instructions given in the study
6. Psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
SNAP-IV teacher form scores in ORADUR®-Methylphenidate | 24 months
  Change from baseline of Swanson, Nolan, and Pelham-IV (SNAP-IV) teacher form scores

SECONDARY OUTCOMES:
SNAP-IV parent form scores in ORADUR®-Methylphenidate | 24 months
  Change from baseline of SNAP-IV parent form scores
Remission rate in ORADUR®-Methylphenidate | 24 months
  Remission rate as assessed by SNAP-IV teacher form and SNAP-IV parent form
Conners' Continuous Performance Test (CPT-II) performance in ORADUR®-Methylphenidate | 24 months
  Change from baseline of Conners' Continuous Performance Test (CPT-II) performance results
Diagnostic & Statistical Manual for Mental Disorders-Fifth Edition (DSM-5) diagnosis in ORADUR®-Methylphenidate | 24 months
  Change from baseline (screening period) of Diagnostic & Statistical Manual for Mental Disorders-Fifth Edition (DSM-5) diagnosis. During study period, DSM-5 diagnosis will be performed at each visit. Investigator will check the diagnostic classification, the dianostic criteria sets and the descriptive test of DSM-5 questionnaire and confirm the severity of ADHD based on subject's current condition.
Clinical Global Impression-ADHD-Severity (CGI-S) scores in ORADUR®-Methylphenidate | 24 months
  Change from baseline of Clinical Global Impression-ADHD-Severity (CGI-S) scores
Clinical Global Impression-ADHD-Improvement (CGI-I) scores in ORADUR®-Methylphenidate | 24 months
  Change from baseline of Clinical Global Impression-ADHD-Improvement (CGI-I) scores
Computerized Cambridge Neuropsychological Test Automated Battery (CANTAB) performance in ORADUR®-Methylphenidate | 24 months
  Change from baseline of Computerized Cambridge Neuropsychological Test Automated Battery (CANTAB) performance result (at National Taiwan University Hospital, NTUH, only)
Treatment compliance in ORADUR®-Methylphenidate | 24 months
  Evaluate the treatment compliance during study period. Compliance will be assessed by the result of drug accountability and presented by the missing dose rate.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Lin, Study Director — Orient pharma
Locations (3):
- Taiwan (3):
  - Chang Gung Medical Foundation- Chiayi Branch, Chiayi City
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation- Linkuo Branch, Taoyuan District